CLINICAL TRIAL: NCT05914701
Title: Efficacy and Safety of Letermovir for Secondary Prophylaxis of Cytomegalovirus Infection After HLA-haploidentical Hematopoietic Stem Cell Transplantation
Brief Title: Secondary Prophylaxis of CMV Infection Using Letermovir After HID-HSCT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-CMV-SP-01
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: To Evaluate the Efficacy and Safety of Secondary Prophylaxis of CMV Reactivation
MeSH Terms: interventions — letermovir

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment arm (Experimental)
  Interventions: Drug: Letermovir for secondary prophylaxis

INTERVENTIONS:
Drug: Letermovir for secondary prophylaxis — For enrolled patients, Letermovir would be administered at a dose of 480 mg per day (or 240 mg per day in patients taking cyclosporine). The regimen duration of dosing was approximately 120 days or 16 weeks. Or physicians could adjust regimen duration according to the CMV infection risk factors.
  Other Names: secondary prophylaxis of CMV reactivation

SUMMARY:
To evaluate the efficacy and safety of secondary prophylaxis of CMV reactivation, clinically significant CMV infection with oral letermovir in Chinese haplo-HSCT patients, as well as treatment-related mortality, all-cause mortality and QoL after transplantation. For enrolled patients, Letermovir would be administered at a dose of 480 mg per day (or 240 mg per day in patients taking cyclosporine). The regimen duration of dosing was approximately 120 days or 16 weeks. Or physicians could adjust regimen duration according to the CMV infection risk factors.

ELIGIBILITY:
Inclusion Criteria:

- (1) Underwent HLA-haploidentical donor HSCT, after at least 1 treated CMV episode since transplant in patients who did not receive primary prophylaxis.

(2) Age elder than or equal to 18 years; (3) Informed consent may be signed by themselves. (4) HIV negative, HBV, HCV negative; (5) Informed consent must be signed before the start of the study procedures, and informed consent must be signed by the patient himself or his immediate family. Considering the patient 's condition, if the patient' s signature is unfavorable for disease treatment, the informed consent form should be signed by the legal guardian or the patient 's immediate family member

Exclusion Criteria:

* (1) received a previous allogeneic HSCT; (2) has evidence of CMV viremia from a central or local laboratory, or CMV end-organ disease within one week prior to enrollment; (3) received within 30 days prior to screening or plans to receive during the study any of the following: cidofovir, or any investigational anti-CMV therapy or biological agent; (4) has severe hepatic insufficiency (defined as Child-Pugh Class C; (5) has serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 5 xthe upper limit of normal (ULN) or serum total bilirubin > 2.5 x ULN.

  (6) has end-stage renal impairment with a creatinine clearance less than 10 mL/min.

  (7) has both moderate hepatic insufficiency AND moderate renal insufficiency; (8) Uncontrolled infection at enrollment; (9) requires mechanical ventilation or is hemodynamically unstable at the time of enrollment; (10) has documented positive results for human immunodeficiency virus antibody (HIVAb), hepatitis C virus antibody (HCV-Ab) with detectable HCV RNA, or hepatitis B surface antigen (HBsAg) within 90 days prior to enrollments; (11) has active solid tumor malignancies with the exception of localized basal cell or squamous cell skin cancer or the condition under treatment (e.g., lymphomas).

  (12) Suffering from mental disorders or other conditions and unable to cooperate with the requirements of study treatment and monitoring; (13) unable or unwilling to sign the consent form; (14) pregnant or lactating women; (15) patients with other special conditions assessed as unqualified by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of CMV reactivation and CMV infection | 1 year after letermovir administration
  The incidence of peripheral blood cytomegalovirus activation and confirmed clinically significant CMV infection occurred within 1 year after treatment; if the patient terminated letemovir treatment for any reason after treatment, or clinical data loss occurred within 1 year, it was also included in the primary endpoint event.